CLINICAL TRIAL: NCT02237287
Title: Combination of Taliderm® and VAC for Treatment of Pressure Ulcers - a Pilot Study
Brief Title: Combination of Taliderm® and Vacuum-assisted Closure (VAC) for Treatment of Pressure Ulcers
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Open label study part reduced from n=10 to n=6 because of insufficient number of patients under antiaggregation.
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Marine Polymer Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010-MD-0007
Record Dates: First submitted 2014-08-18; First posted 2014-09-11 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Wounds; Pressure Ulcer
MeSH Terms: conditions — Wounds and Injuries; Pressure Ulcer | interventions — Bandages

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- wound dressing with VAC (Sham Comparator): After wound debridement wounds are treated for 2 weeks with VAC dressing alone
  Interventions: Procedure: wound dressing with VAC
- wound dressing with VAC and sNAG under Antiaggregation (Other): In patients being under antiaggregation with Aspirin® 100mg daily, after wound debridement wounds are treated with VAC and sNAG
  Interventions: Other: wound dressing with VAC and sNAG without antiaggregation; Procedure: wound dressing with VAC; Drug: wound dressing with VAC and sNAG under Antiaggregation
- wound dressing with VAC and sNAG without antiaggregation (Experimental): In patients NOT being under antiaggregation, after wound debridement wounds are treated with VAC and sNAG
  Interventions: Other: wound dressing with VAC and sNAG without antiaggregation; Procedure: wound dressing with VAC

INTERVENTIONS:
Other: wound dressing with VAC and sNAG without antiaggregation
  Arms: wound dressing with VAC and sNAG under Antiaggregation; wound dressing with VAC and sNAG without antiaggregation
Procedure: wound dressing with VAC
Drug: wound dressing with VAC and sNAG under Antiaggregation
  Arms: wound dressing with VAC and sNAG under Antiaggregation

SUMMARY:
Background: The wound healing promoting effect of negative wound pressure therapies (NWPT) takes place at the wound foam interface. Implementation of bioactive substances at this site represents a major research area for the development of future NWPT devices.

Methods: Wound healing kinetics of pressure ulcers treated by vacuum assisted closure devices with or without the implementation of a thin interface of poly-N-acetyl glucosamine nanofibers (sNAG) was studied in a prospective randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Ischial/sacral Pressure ulcer between 4 and 15cm diameter
* Greater than or equal to 18 years of age
* Ability to obtain informed consent

Exclusion Criteria:

* Connective tissue disorders
* Immunosuppression, Hemodialysis, Steroids
* Pregnancy
* Sepsis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | up to 1 year
Wound surface area increase, respectively decrease as a measure of the effect of the studied devices on pressure ulcer healing | up to 1 year

SECONDARY OUTCOMES:
Wound Healing characteristics | up to 1 year
  Evaluation of granulation tissue formation in study groups
Wound Healing characteristics | up to 1 year
  Evaluation of wound epithelialization in study groups
Wound Healing characteristics | up to 1 year
  Evaluation of wound contraction in study groups

CONTACTS AND LOCATIONS:
Overall Officials: Dirk J. Schaefer, Prof.Dr., Study Director — University Hospital, Basel, Switzerland
Locations (2):
- Switzerland (2):
  - University Hospital Basel, Basel
  - Swiss Paraplegic Centre Nottwil, Nottwil